CLINICAL TRIAL: NCT06864494
Title: L-PGDS (Lipocalin Type- Prostaglandin) Quantification in Genital, Blood and Urine Samples From Adenomyosis Patients Compared to 2 Control Groups.
Brief Title: Determination of Lipocalin Type-prostaglandin (L-PGDS) in Blood, Urine, Vaginal Samples and Endometrial Ablation by Enzyme-linked Immunosorbent Assay
Acronym: ADENO-L
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2024-1/SH01
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Adenomyosis; Endometriosis
Keywords: lipocalin-Type Prostaglandin D2 Synthase
MeSH Terms: conditions — Adenomyosis; Endometriosis | interventions — Endometrial Ablation Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swabs, endometrial ablation samples, urine, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with adenomyosis (Adenomyosis +)
  Interventions: Procedure: Endometrial ablation
- Patients with an endometrial pathology other than adenomyosis (Adenomyosis -)
  Interventions: Procedure: Endometrial ablation
- Patients without uterine pathology (control)

INTERVENTIONS:
Procedure: Endometrial ablation — Performed using a transfer catheter (used for embryo transfers) positioned at the level of the internal cervical orifice in the uterine cavity. Five ml of saline will be injected and collected in a dry tube
  Groups: Patients with adenomyosis (Adenomyosis +); Patients with an endometrial pathology other than adenomyosis (Adenomyosis -)

SUMMARY:
Prostaglandin D2 (PGD2) has anti-inflammatory activity, particularly via Lipocalin type-prostaglandin (L-PGDS). L-PGDS has been studied in pathologies such as sleep apnea, rheumatoid arthritis, asthma and allergic phenomena, but never in adenomyosis. Adenomyosis is a estrogen-dependent multifactorial pathology whose pathophysiology is still poorly defined. This hyperestrogenism causes chronic inflammation, particularly via the activation of the prostaglandin H2 (PGH2) signaling pathway. This would lead to the excess production of prostaglandins E2 (PGE2) and F2a (PGF2a) and the decrease of PGD2 and therefore of L-PGDS, leading to the proliferation of endometrial cells in the myometrium by the epithelial-mesenchymal transition via aromatase. A preliminary study comparing the expression of L-PGDS found a significant decrease in L-PGDS in the uterus of women with adenomyosis lesions versus healthy controls. However, during this study, some information was not collected, including the patients' symptoms, preoperative radiological data and surgical indication. The study authors hypothesize that L-PGDS could be a potential tissue and circulating diagnostic marker of adenomyosis in its early stages. L-PGDS appears to be a good candidate to aid in the diagnosis of adenomyosis via a minimally invasive assay for patients (blood or urine).

ELIGIBILITY:
Inclusion Criteria:

Common inclusion criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Adenomyosis + group:

* Female.
* Aged 40 (≥) to 55 (≤) years.
* Multiparous.
* Non-menopausal.
* Having an indication for a total inter-ovarian hysterectomy (excluding oncology).
* Suffering from adenomyosis.

Adenomyosis - group:

* Female.
* Aged 40 (≥) to 55 (≤) years.
* Multiparous.
* Non-menopausal.
* Having an indication for a total inter-ovarian hysterectomy (excluding oncology).
* Suffering from a functional pathology other than adenomyosis.

Control Group:

* Female.
* Aged 18 (≥) to 43 (≤) years.
* Nulliparous.
* Asymptomatic: absence of menometrorrhagia and pelvic pain.
* Support at the medically assisted procreation (MAP) center of the Nîmes University Hospital for male or idiopathic infertility.
* Indication to perform an endovaginal ultrasound as part of MAP management.
* Absence of uterine pathology visualized on endovaginal ultrasound.

Exclusion Criteria:

* History of autoinflammatory or autoimmune disease.
* History of atopic or asthmatic conditions.
* History of sleep apnea syndrome.
* Chronic or acute renal failure.
* Liver failure
* History of active neoplasia or cancer.
* Presence of a functional-looking ovarian cyst on imaging (endovaginal ultrasound and/or pelvic MRI).
* Taking nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroids, or aspirin in the 15 days prior to L-PGDS concentration measurement
* Undergoing estrogen-progestin hormonal contraception.

Adenomyosis groups:

- Contraindication to MRI.

Control Group:

- Endovaginal ultrasound refused by the patient.

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Multiparous, non-menopausal patients aged between 40 and 55 consulting the gynecology-obstetrics department of the CHU de Nîmes for menometrorrhagia and/or pelvic pain and having an indication for total inter-ovarian hysterectomy plus healthy controls aged between 18 and 43, nulliparous, without uterine pathologies treated at the Nîmes University Hospital's assisted reproduction center for male or idiopathic infertility.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of L-PGDS in vaginal swabs between groups | Day 0
  Assessed with immunoenzymatic ELISA (µg/ml)
Concentration of L-PGDS in endometrial ablation sample in Adenomyosis - and + groups | Day 0
  Assessed with immunoenzymatic ELISA (µg/ml) Day 0

SECONDARY OUTCOMES:
Concentration of L-PGDS in blood between groups | Day 0
  Assessed with immunoenzymatic ELISA (µg/ml) Day 0
Concentration of L-PGDS in blood between groups | 7 weeks (range 6 to 8 weeks)
  Assessed with immunoenzymatic ELISA (µg/ml) Day 0
Concentration of L-PGDS in urine between groups | Day 0
  Assessed with immunoenzymatic ELISA (µg/ml) Day 0
Concentration of L-PGDS in urine between groups | 7 weeks (range 6 to 8 weeks)
  Assessed with immunoenzymatic ELISA (µg/ml) Day 0
Adenomyosis severity grade | Day 0
  Measured by MRI. Severity grade: minimal (<25%), moderate (25-50%) or severe (>50%) uterine involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie HUBERLANT, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No